CLINICAL TRIAL: NCT02755402
Title: Impact of an Accelerated Pre-treatment Evaluation on Linkage-to-care and Linkage-to-treatment for HCV Infected Persons Who Inject Drugs
Brief Title: Accelerated Pre-treatment Evaluation for HCV Infected Persons Who Inject Drugs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Gilead Sciences (Industry); Cepheid (Industry)
Responsible Party: Principal Investigator, Valérie Martel-Laferrière, Medical microbiologist, Centre hospitalier de l'Université de Montréal (CHUM)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IN-CA-337-2100
Record Dates: First submitted 2016-04-20; First posted 2016-04-28 (Estimated); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Hepatitis C; Intravenous Drug Users
MeSH Terms: conditions — Hepatitis C

ARMS (1):
- Rapid evaluation (Experimental): Transient elastography, Xpert HCV Viral load, medical and nurse visits
  Interventions: Device: Xpert HCV Viral load; Device: Transient elastography

INTERVENTIONS:
Device: Xpert HCV Viral load — HCV viral load testing
Device: Transient elastography — Evaluation of liver fibrosis

SUMMARY:
Persons who inject drugs (PWID) are overrepresented among hepatitis C infected patients, but underrepresented among those who are treated, despite many studies showing that treatment is feasible and effective in this population.

The hepatitis C diagnosis and pre-treatment evaluation are multistep processes. Every step is a potential occasion for disengagement and loss to follow-up. This is especially true with hard-to-reach populations such as PWID in whom competing needs are numerous and psychosocial situation can change rapidly.

By using new technologies that can quickly provide clinical results, like Xpert HCV Viral Load (Cepheid) and transient elastography (fibroscan), a provider could determine if a patient needs treatment rapidly or not on the day of the initial visit.

The aim of this study is to explore whether an accelerated pre-treatment evaluation can result in an improved linkage-to-care (defined as linkage to health care, addiction or social services) and, eventually, linkage-to-treatment among PWID.

DETAILED DESCRIPTION:
This is a non-randomized, open-label study that aims to include HCV-infected patients who inject drugs and who do not know their treatment eligibility status. A total of 200 patients will be evaluated using our rapid evaluation protocol, which will include basic blood tests, viral load measurement using Cepheid's Xpert® HCV Viral Load technique (which will be controlled at the same time by COBAS® AmpliPrep/ COBAS® TaqMan® HCV Quantitative Test, version 2.0 (Roche), available at the CHUM and approved by Health Canada), a liver fibrosis assessment and HCV genotyping. The results of the basic tests, viral load tests and FibroScan® test will be available on the same day as the patient's visit and will allow the investigator to determine straightaway whether or not the patient is treatable based on the RAMQ's reimbursement criteria at the time of the study.

If the patient is treatable, once the genotype result has been obtained, the most appropriate treatment for their medical condition, degree of liver fibrosis and genotype will be prescribed. There will be no other visits between the initial visit and the treatment initiation visit. The patient will be given an appointment for the treatment initiation visit once the medication has been approved by the RAMQ or the patient's private insurer. The patient will be seen again at weeks 2 and 4 of treatment, at the end of treatment (usually week 12), then 12, 24 and 36 weeks post-treatment.

If the patient is not treatable, he/she will be referred to the CHUM Addiction Medicine Clinic or the UHRESS (if HIV-coinfected status) for management, which will include longitudinal follow-up of his HCV and substance abuse. The patient will be seen again at 6 months and 1 year to determine whether or not there has been linkage-to-care, initiation of opioid substitution therapy if indicated and if the patient has reduced his injection drug use.

If an untreatable patient becomes treatable during follow-up, treatment will be offered.

At the same time, we will review the records of patients seen at the CHUM Addiction Medicine Clinic between October 2014 and June 2016 who meet the inclusion criteria for the study cohort and the RAMQ's treatment eligibility criteria. This cohort will be used as an historical cohort to determine the rate of linkage to treatment with the standard pre-treatment evaluation protocol.

ELIGIBILITY:
Inclusion Criteria:

* Person who inject drugs, defined as having injected in the past year
* Able to give an informed consent
* Unknown treatment eligibility status

Exclusion Criteria:

* Patients actively engaged in HCV follow up
* Patients visibly intoxicated at initial study visit
* Pregnant or breastfeeding women
* Pacemaker.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2021-05 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who initiate treatment after first visit | 1 year
  Proportion of patients who initiate treatment among those who are treatment-eligible based on Quebec's treatment reimbursement guidelines following the accelerated intervention and comparison with historical controls

SECONDARY OUTCOMES:
Proportion of patients who attend at least two visits in 6 months | 6 months
  To compare linkage-to-care proportion at one year of treated PWID with untreated PWID at one year.
Proportion of patients who initiate opioid substitution therapy during follow-up | 6 months
  To compare opioid substitution therapy initiation rates at one year of treated and untreated PWID.
Difference in number of injection between the month prior to study entry and the last month of follow-up | 6 months
  To compare drug use reduction during the study period of treated PWID with untreated PWID at one year.
Sustained virological response (undetectable HCV viral load 12 weeks post-end-of-treatment | 12 weeks post-treatment
  To compare proportion of treated patients who achieved SVR12 with historical controls treated in phase III trials.
Proportion of patients with a re-infection within six months of end-of-treatment | 6 months post-treatment
  To evaluate rapid re-infection rates (<6 months) of patients who achieve end-of-treatment undetectability.
Difference in HCV viral load results between techniques | At enrollment
  To compare Xpert HCV Viral Load® (Cepheid) viral loads results to HCV RealTime® (Abbott) results.
Recontact of initially untreatable patients | 1 year
  To determine the proportion of patients who change from untreatable to treatable that can be successfully recontacted and linked to care among patients initially classified as untreatable
Treatment of initially untreatable patients | 1 year
  To determine the proportion of patients who will initiate HCV treatment among those who were initially classified as untreable.

CONTACTS AND LOCATIONS:
Overall Officials: Valérie Martel-Laferrière, MD, MSc, Principal Investigator — CRCHUM
Locations (1):
- Centre hospitalier de l'Université de Montréal, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Martel-Laferriere V, Brissette S, Wartelle-Bladou C, Juteau LC, Popa M, Goyer ME, Bruneau J. Impact of an Accelerated Pretreatment Evaluation on Linkage-to-Care for Hepatitis C-infected Persons Who Inject Drugs. Subst Abuse. 2022 Aug 12;16:11782218221119068. doi: 10.1177/11782218221119068. eCollection 2022. PMID 35990750